CLINICAL TRIAL: NCT01105247
Title: A Phase 1b/2 Fixed-dose Study of Bruton's Tyrosine Kinase (Btk) Inhibitor, PCI-32765, in Chronic Lymphocytic Leukemia
Brief Title: Safety of PCI-32765 in Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1102-CA; PCI-32765 (Other: Pharmacyclics)
Record Dates: First submitted 2010-04-13; First posted 2010-04-16 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-02

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: PCI-32765; Lymphoma, B-Cell; Leukemia, Lymphoid; Leukemia, B-Cell; Bruton's Tyrosine Kinase
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Leukemia, Lymphoid; Leukemia, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PCI-32765 (Experimental)
  Interventions: Drug: PCI-32765

INTERVENTIONS:
Drug: PCI-32765 — 420 mg daily or 840 mg daily

SUMMARY:
The purpose of this study is to establish the safety and efficacy of orally administered PCI-32765 in patients with chronic lymphocytic leukemia/small lymphocytic lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. FOR TREATMENT-NAIVE GROUP ONLY: Men and women ≥ 65 years of age with confirmed diagnosis of CLL/SLL, who require treatment per NCI or International Working Group guidelines 15-18
2. FOR RELAPSED/REFRACTORY GROUP ONLY: Men and women ≥ 18 years of age with a confirmed diagnosis of relapsed/refractory CLL/SLL following previous therapy(ie, failed ≥ 2 previous treatments for CLL/SLL and at least 1 regimen had to have had a purine analog [eg, fludarabine] for subjects with CLL)
3. FOR HIGH-RISK RELAPSED/ REFRACTORYGROUP ONLY: Men and women ≥ 18 years of age with a confirmed diagnosis of relapsed/refractory CLL/SLL with suboptimal response to chemoimmunotherapy, defined as progression of disease within 24 months of initiation of a regimen containing at least a nucleoside analogue or bendamustine in combination with a monoclonal antibody or failure to respond to such a regimen. (Note: a minimum of 2 cycles of chemoimmunotherapy required for eligibility)
4. ECOG performance status of ≤ 2
5. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty

Exclusion Criteria:

1. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for at least 2 years or which will not limit survival to < 2 years
2. Any immunotherapy, chemotherapy, radiotherapy, or experimental therapy within 4 weeks before first dose of study drug (corticosteroids for disease-related symptoms allowed but require 1-week washout before study drug administration)
3. Central nervous system (CNS) involvement by lymphoma
4. Major surgery within 4 weeks before first dose of study drug
5. Concomitant use of medicines known to cause QT prolongation or torsades de pointes
6. Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree AV block type II, 3rd degree block, bradycardia, and QTc > 470 msec
7. Lactating or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danelle James, M.D., M.A.S, Study Director — Pharmacyclics LLC.
Locations (10):
- United States (10):
  - Stanford University School of Medicine, Stanford, California
  - New York Presbyterian Hosptial Cornell Med Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Sarah Cannon, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - University of Vermont and Fletcher Allen Health Care, Burlington, Vermont
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Yakima Valley Memorial, Yakima, Washington

REFERENCES:
- [Derived] Byrd JC, Furman RR, Coutre SE, Flinn IW, Burger JA, Blum K, Sharman JP, Wierda W, Zhao W, Heerema NA, Luan Y, Liu EA, Dean JP, O'Brien S. Ibrutinib Treatment for First-Line and Relapsed/Refractory Chronic Lymphocytic Leukemia: Final Analysis of the Pivotal Phase Ib/II PCYC-1102 Study. Clin Cancer Res. 2020 Aug 1;26(15):3918-3927. doi: 10.1158/1078-0432.CCR-19-2856. Epub 2020 Mar 24. PMID 32209572
- [Derived] Coutre SE, Byrd JC, Hillmen P, Barrientos JC, Barr PM, Devereux S, Robak T, Kipps TJ, Schuh A, Moreno C, Furman RR, Burger JA, O'Dwyer M, Ghia P, Valentino R, Chang S, Dean JP, James DF, O'Brien SM. Long-term safety of single-agent ibrutinib in patients with chronic lymphocytic leukemia in 3 pivotal studies. Blood Adv. 2019 Jun 25;3(12):1799-1807. doi: 10.1182/bloodadvances.2018028761. PMID 31196847
- [Derived] O'Brien SM, Jaglowski S, Byrd JC, Bannerji R, Blum KA, Fox CP, Furman RR, Hillmen P, Kipps TJ, Montillo M, Sharman J, Suzuki S, James DF, Chu AD, Coutre SE. Prognostic Factors for Complete Response to Ibrutinib in Patients With Chronic Lymphocytic Leukemia: A Pooled Analysis of 2 Clinical Trials. JAMA Oncol. 2018 May 1;4(5):712-716. doi: 10.1001/jamaoncol.2017.5604. PMID 29470582
- [Derived] O'Brien S, Furman RR, Coutre S, Flinn IW, Burger JA, Blum K, Sharman J, Wierda W, Jones J, Zhao W, Heerema NA, Johnson AJ, Luan Y, James DF, Chu AD, Byrd JC. Single-agent ibrutinib in treatment-naive and relapsed/refractory chronic lymphocytic leukemia: a 5-year experience. Blood. 2018 Apr 26;131(17):1910-1919. doi: 10.1182/blood-2017-10-810044. Epub 2018 Feb 2. PMID 29437592
- [Derived] Fraietta JA, Beckwith KA, Patel PR, Ruella M, Zheng Z, Barrett DM, Lacey SF, Melenhorst JJ, McGettigan SE, Cook DR, Zhang C, Xu J, Do P, Hulitt J, Kudchodkar SB, Cogdill AP, Gill S, Porter DL, Woyach JA, Long M, Johnson AJ, Maddocks K, Muthusamy N, Levine BL, June CH, Byrd JC, Maus MV. Ibrutinib enhances chimeric antigen receptor T-cell engraftment and efficacy in leukemia. Blood. 2016 Mar 3;127(9):1117-27. doi: 10.1182/blood-2015-11-679134. Epub 2016 Jan 26. PMID 26813675
- [Derived] Maddocks KJ, Ruppert AS, Lozanski G, Heerema NA, Zhao W, Abruzzo L, Lozanski A, Davis M, Gordon A, Smith LL, Mantel R, Jones JA, Flynn JM, Jaglowski SM, Andritsos LA, Awan F, Blum KA, Grever MR, Johnson AJ, Byrd JC, Woyach JA. Etiology of Ibrutinib Therapy Discontinuation and Outcomes in Patients With Chronic Lymphocytic Leukemia. JAMA Oncol. 2015 Apr;1(1):80-7. doi: 10.1001/jamaoncol.2014.218. PMID 26182309
- [Derived] de Jong J, Sukbuntherng J, Skee D, Murphy J, O'Brien S, Byrd JC, James D, Hellemans P, Loury DJ, Jiao J, Chauhan V, Mannaert E. The effect of food on the pharmacokinetics of oral ibrutinib in healthy participants and patients with chronic lymphocytic leukemia. Cancer Chemother Pharmacol. 2015 May;75(5):907-16. doi: 10.1007/s00280-015-2708-9. Epub 2015 Feb 28. PMID 25724156
- [Derived] Marostica E, Sukbuntherng J, Loury D, de Jong J, de Trixhe XW, Vermeulen A, De Nicolao G, O'Brien S, Byrd JC, Advani R, McGreivy J, Poggesi I. Population pharmacokinetic model of ibrutinib, a Bruton tyrosine kinase inhibitor, in patients with B cell malignancies. Cancer Chemother Pharmacol. 2015 Jan;75(1):111-21. doi: 10.1007/s00280-014-2617-3. Epub 2014 Nov 8. PMID 25381051
- [Derived] O'Brien S, Furman RR, Coutre SE, Sharman JP, Burger JA, Blum KA, Grant B, Richards DA, Coleman M, Wierda WG, Jones JA, Zhao W, Heerema NA, Johnson AJ, Izumi R, Hamdy A, Chang BY, Graef T, Clow F, Buggy JJ, James DF, Byrd JC. Ibrutinib as initial therapy for elderly patients with chronic lymphocytic leukaemia or small lymphocytic lymphoma: an open-label, multicentre, phase 1b/2 trial. Lancet Oncol. 2014 Jan;15(1):48-58. doi: 10.1016/S1470-2045(13)70513-8. Epub 2013 Dec 10. PMID 24332241
- [Derived] Dubovsky JA, Beckwith KA, Natarajan G, Woyach JA, Jaglowski S, Zhong Y, Hessler JD, Liu TM, Chang BY, Larkin KM, Stefanovski MR, Chappell DL, Frissora FW, Smith LL, Smucker KA, Flynn JM, Jones JA, Andritsos LA, Maddocks K, Lehman AM, Furman R, Sharman J, Mishra A, Caligiuri MA, Satoskar AR, Buggy JJ, Muthusamy N, Johnson AJ, Byrd JC. Ibrutinib is an irreversible molecular inhibitor of ITK driving a Th1-selective pressure in T lymphocytes. Blood. 2013 Oct 10;122(15):2539-49. doi: 10.1182/blood-2013-06-507947. Epub 2013 Jul 25. PMID 23886836
- [Derived] Byrd JC, Furman RR, Coutre SE, Flinn IW, Burger JA, Blum KA, Grant B, Sharman JP, Coleman M, Wierda WG, Jones JA, Zhao W, Heerema NA, Johnson AJ, Sukbuntherng J, Chang BY, Clow F, Hedrick E, Buggy JJ, James DF, O'Brien S. Targeting BTK with ibrutinib in relapsed chronic lymphocytic leukemia. N Engl J Med. 2013 Jul 4;369(1):32-42. doi: 10.1056/NEJMoa1215637. Epub 2013 Jun 19. PMID 23782158
- See also: Related Info — http://www.pharmacyclics.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There are total 133 subjects enrolled however one subject never received treatment. Therefore, number of subjects "Started" the study is listed as 132 subjects.
Groups:
- Food Effect Cohort: PCI-32765: 420 mg daily
Period: Overall Study
Arm/Group | PCI-32765 | Food Effect Cohort
Started | 116 | 16
Completed | 79 | 16
Not Completed | 37 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCI-32765 | Food Effect Cohort | Total
Number analyzed (Participants) | 116 | 16 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 9 | 51
  >=65 years | 74 | 7 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 2 | 34
  Male | 84 | 14 | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: Number of participants who had experienced at least one treatment emergent AEs.
Time Frame: From first dose to within 30 days of last dose of PCI-32765
Measure: Number; unit: Participants
Groups:
- Food Effect: Food-Effect Relapsed/Refractory participants received PCI-32765 420 mg daily
Arm/Group | PCI-32765 | Food Effect
Number analyzed (Participants) | 116 | 16
Participants | 116 | 11

2. Secondary Outcome: Food Effect Cohort Assessments
Description: Geometric mean ratio (Fed/Fasted) for PCI-32765 AUClast. The data were collected at 0, 0.5, 1, 2, 4, 6, 24 h post-dose. The AUClast was calculated from 0 up to 24 hours post-dose.
Time Frame: Fed was assessed on either Day 8 or Day 15 and Fasted was assessed on the remaining day as cross-over design.
Population: Note: 16 subjects were participated in food effect cohort. However, the PK parameters for 1 subject under Fasted treatment period cannot be reliably estimated. The data for this subject were excluded from Fed/Fasted comparison.
Measure: Number (90% Confidence Interval)
Arm/Group | Food Effect Cohort
Number analyzed (Participants) | 15
Value | 1.65 [1.23 to 2.19]

3. Secondary Outcome: Progression Free Survival Rate at 24 Months
Description: Criteria for progression are as outlined in the IWCLL 2008 criteria (Hallek 2008) and as assessed by investigator, e.g. progression defined as a 50% increase in lymph node size.
Time Frame: The median follow-up time for all treated patients are 21 month, range (0.7 month, 29 months).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Treatment Naive; Relapsed/ Refractory: PCI-32765: 420 mg daily or 840 mg daily
- Food- Effect: Food-Effect Relapsed/refractory participants received PCI-32765 420 mg daily
Arm/Group | Treatment Naive | Relapsed/ Refractory | Food- Effect
Number analyzed (Participants) | 31 | 85 | 16
Percentage of Participants | 96.3 [76.5 to 99.5] | 73.6 [60.2 to 83.1] | NA [NA to NA] — There was no PD or death occurred in this arm.

4. Secondary Outcome: Percentage of Participants Achieving Response
Description: Response criteria are as outlined in the IWCLL 2008 criteria (Hallek 2008) and as assessed by investigator, e.g. response requires 50% reduction in lymph node size.
Time Frame: The median follow-up time for all treated patients are 21 month, range (0.7 month, 29 months).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment Naive | Relapsed/ Refractory | Food Effect
Number analyzed (Participants) | 31 | 85 | 16
Percentage of Participants | 71 [52 to 85.8] | 75.3 [64.7 to 84] | 56.3 [29.9 to 80.2]

ADVERSE EVENTS:
Groups:
- Food Effect: PCI-32765: 420 mg daily
Arm/Group | PCI-32765 | Food Effect
Serious Adverse Events (participants affected / at risk) | 61/116 | 7/16
Other Adverse Events (participants affected / at risk) | 116/116 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCI-32765 (N=116) | Food Effect (N=16)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
Splenomegaly (Blood and lymphatic system disorders) | 2 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 11 | 4
Bacteraemia (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 4 | 0
Sinusitis (Infections and infestations) | 4 | 0
Sepsis (Infections and infestations) | 3 | 0
Clostridial infection (Infections and infestations) | 2 | 0
Pneumonia viral (Infections and infestations) | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Citrobacter infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 1 | 0
Joint abscess (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0
Pneumonia cryptococcal (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral Infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukostasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PCI-32765 (N=116) | Food Effect (N=16)
Anaemia (Blood and lymphatic system disorders) | 19 | 0
Neutropenia (Blood and lymphatic system disorders) | 16 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 15 | 0
Dry eye (Eye disorders) | 11 | 0
Cataract (Eye disorders) | 6 | 0
Conjunctivitis (Eye disorders) | 6 | 1
Constipation (Gastrointestinal disorders) | 25 | 1
Dyspepsia (Gastrointestinal disorders) | 17 | 0
Stomatitis (Gastrointestinal disorders) | 16 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 1
Dry mouth (Gastrointestinal disorders) | 7 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 6 | 0
Fatigue (General disorders) | 38 | 4
Oedema peripheral (General disorders) | 33 | 1
Chills (General disorders) | 14 | 3
Malaise (General disorders) | 9 | 1
Pain (General disorders) | 6 | 1
Allergy to arthropod bite (Immune system disorders) | 7 | 0
Bronchitis (Infections and infestations) | 9 | 0
Nasopharyngitis (Infections and infestations) | 8 | 0
Fungal infection (Infections and infestations) | 6 | 1
Gastroenteritis viral (Infections and infestations) | 6 | 0
Oral herpes (Infections and infestations) | 6 | 0
Contusion (Injury, poisoning and procedural complications) | 22 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 8 | 2
Weight decreased (Investigations) | 8 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 6 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 0
Anxiety (Psychiatric disorders) | 15 | 1
Insomnia (Psychiatric disorders) | 14 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 17 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 14 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 11 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 8 | 0
Erythema (Skin and subcutaneous tissue disorders) | 8 | 0
Rash (Skin and subcutaneous tissue disorders) | 8 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 7 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 | 0
Hypotension (Vascular disorders) | 8 | 0
Vision Blurred (Eye disorders) | 6 | 1
Conjuctival hyperaemia (Eye disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 65 | 11
Vomiting (Gastrointestinal disorders) | 22 | 11
Food poisoning (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 31 | 2
Abdominal distension (Gastrointestinal disorders) | 5 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Oral mucosal blistering (Gastrointestinal disorders) | 1 | 1
Early satiety (General disorders) | 3 | 1
Injection site haematoma (General disorders) | 0 | 1
Hypogammaglobulinaemia (General disorders) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 37 | 4
Cellulitis (Infections and infestations) | 7 | 1
Folliculitis (Infections and infestations) | 5 | 1
Furuncle (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 3 | 1
Urinary track infection (Infections and infestations) | 14 | 1
Laceration (Injury, poisoning and procedural complications) | 7 | 2
Excoriation (Injury, poisoning and procedural complications) | 2 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 1
Blood urea increased (Investigations) | 2 | 1
Cardiac murmur (Investigations) | 4 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 1
Headache (Nervous system disorders) | 22 | 4
Depression (Psychiatric disorders) | 4 | 1
Urinary retention (Renal and urinary disorders) | 3 | 2
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 4 | 2
Blood blister (Skin and subcutaneous tissue disorders) | 2 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 2
Blister (Skin and subcutaneous tissue disorders) | 1 | 1
Pityriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Pseudoporphyria (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 5 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 27 | 2
Lymphoedema (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No